CLINICAL TRIAL: NCT00858364
Title: A Randomized, Double-blind, Placebo-controlled Study to Evaluate the Long-term Safety and Efficacy of Darbepoetin Alfa Administered at 500 µg Once-Every-3-Weeks in Anemic Subjects With Advanced Stage Non-small Cell Lung Cancer Receiving Multi-cycle Chemotherapy
Brief Title: Anemia Treatment for Advanced Non-Small Cell Lung Cancer (NSCLC) Patients Receiving Chemotherapy
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 20070782; 2007-005792-34 (EudraCT Number)
Record Dates: First submitted 2009-03-05; First posted 2009-03-09 (Estimated); Results first posted 2018-07-06 (Actual); Last update posted 2022-11-30 (Actual); Status verified 2022-11

CONDITIONS: Non-Small Cell Lung Cancer; Anemia; Cancer; Lung Cancer
Keywords: darbepoetin alfa; non-small cell lung cancer; Aranesp; chemotherapy; chemotherapy induce anemia; advanced lung cancer; malignant pleural effusion; metastatic lung cancer; NSCLC; anemia; lung cancer; pleural effusion; Stage IIIB lung cancer; Stage IV lung cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Anemia; Neoplasms; Lung Neoplasms; Pleural Effusion, Malignant; Pleural Effusion | interventions — Darbepoetin alfa

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Participants received placebo once every 3 weeks (Q3W) administered subcutaneously until 3 weeks after the completion of chemotherapy or upon determination of disease progression, whichever occurred first.
  Interventions: Drug: Placebo
- Darbepoetin alfa (Experimental): Participants received darbepoetin alfa 500 µg once every 3 weeks (Q3W) administered subcutaneously until 3 weeks after the completion of chemotherapy or upon determination of disease progression, whichever occurred first.
  Interventions: Drug: Darbepoetin alfa

INTERVENTIONS:
Drug: Darbepoetin alfa — Administered subcutaneously once every 3 weeks
  Other Names: Aranesp®
  Arms: Darbepoetin alfa
Drug: Placebo — Administered subcutaneously once every 3 weeks
  Arms: Placebo

SUMMARY:
This is a study in patients with chemotherapy induced anemia receiving multi-cycle chemotherapy for the treatment of stage IV non-small cell lung cancer (NSCLC). The primary objective of the study is to demonstrate that overall survival (OS) is not worse in participants on darbepoetin alfa treated to a hemoglobin ceiling of 12.0 g/dL compared to participants treated with placebo.

DETAILED DESCRIPTION:
Oversight Authorities continued: Colombia

ELIGIBILITY:
Inclusion Criteria:

* Subjects with stage IV NSCLC (not recurrent or re-staged).
* Expected to receive at least 2 additional cycles (at least 6 total weeks) of first line myelosuppressive cyclic chemotherapy after randomization. Subjects should not be expected to receive only maintenance chemotherapy.
* Eastern Cooperative Oncology Group performance status of 0 or 1 as assessed within 21 days prior to randomization.
* 18 years of age or older at screening.
* Life expectancy greater than 6 months based on the judgment of the investigator and documented during screening.
* Hemoglobin level less than or equal to 11.0 g/dL as assessed by the local laboratory; sample obtained within 7 days prior to randomization (retest in screening is acceptable).
* Adequate serum folate (greater than or equal to 2 ng/mL) and vitamin B12 (greater than or equal to 200 pg/mL) levels assessed by central laboratory (supplementation and retest acceptable) during screening.
* Subjects must have had a baseline scan (computed tomography [CT], magnetic resonance imaging [MRI], or positron emission tomography-computer tomography [PET/CT]) of the chest to assess disease burden before starting on first line chemotherapy for NSCLC and those images must have been reviewed by the investigator prior to randomization. If the scan was performed more than 28 days prior to randomization, an additional scan must be performed and reviewed by the investigator to confirm that the patient has not progressed before randomization.
* Before any study-specific procedure, the appropriate written informed consent must be obtained from the subject or a legally accepted representative.

Exclusion Criteria:

* Known primary benign or malignant hematologic disorder which can cause anemia.
* History of, or current active cancer other than NSCLC, with the exception of curatively resected non-melanomatous skin cancer, curatively treated cervical carcinoma in situ, or other primary solid tumors curatively treated with no known active disease present and no curative treatment administered for the last 3 years.
* Received any prior adjuvant or neoadjuvant therapy for NSCLC.
* Subjects with a history of brain metastasis.
* Uncontrolled hypertension (systolic blood pressure [BP] > 160 mmHg or diastolic BP > 100 mmHg), or as determined by the investigator during screening.
* History of neutralizing antibody activity to recombinant human erythropoietin (rHuEPO) or darbepoetin alfa.
* Uncontrolled angina, uncontrolled heart failure, or uncontrolled cardiac arrhythmia as determined by the investigator at screening. Subjects with known myocardial infarction within 6 months prior to randomization.
* Subjects with a history of seizure disorder taking anti-seizure medication within 30 days prior to randomization.
* Clinically significant systemic infection or uncontrolled chronic inflammatory disease (eg, rheumatoid arthritis, inflammatory bowel disease) as determined by the investigator during screening.
* Known seropositivity for human immunodeficiency virus (HIV) or diagnosis of acquired immunodeficiency syndrome (AIDS), positive for hepatitis B surface antigen, or seropositive for hepatitis C virus
* History of pure red cell aplasia
* History of deep venous thrombosis or embolic event (eg, pulmonary embolism) within 6 months prior to randomization.
* Transferrin saturation < 20% and ferritin < 50 ng/mL as assessed by the central laboratory during screening. Subjects must have both to be excluded (supplementation and retest acceptable).
* Abnormal renal function (serum creatinine level > 2X upper limit of normal [ULN]) as assessed by the central laboratory during screening.
* Abnormal liver function (total bilirubin > 2X ULN or liver enzymes alanine aminotransferase [ALT] or aspartate aminotransferase [AST] > 2.5X ULN for subjects without liver metastasis or ≥ 5X ULN for subjects with liver metastasis) as assessed by the central laboratory during screening. Subjects with documented Gilbert's Disease may be eligible.
* Received any red blood cell (RBC) transfusion within 28 days prior to randomization.
* Plan to receive any RBC transfusion between randomization and study day 1.
* Known previous treatment failure to erythropoiesis stimulating agents (ESAs) (eg, rHuEPO, darbepoetin alfa).
* ESA therapy within the 28 days prior to randomization.
* Known hypersensitivity to recombinant ESAs or the excipients contained within the investigational product.
* Less than 30 days since receipt of any investigational product or device. Investigational use/receipt of a medicinal product or device that has been approved by the country's local regulatory authority for any indication is permitted.
* Subjects of reproductive potential who are pregnant, breast feeding or not willing to use effective contraceptive precautions during the study and for at least one month after the last dose of investigational product in the judgment of the investigator (including females of childbearing potential who are partners of male subjects).
* Previously randomized to this study.
* Investigator has concerns regarding the ability of the subject to give written informed consent and/or to comply with study procedures (including availability for follow up visits).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2549 (Actual)
Dates: Start 2009-07-17 (Actual); Primary Completion 2017-06-07 (Actual); Study Completion 2017-06-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (482):
- United States (246):
  - Research Site, Anniston, Alabama
  - Research Site, Birmingham, Alabama
  - Research Site, Anchorage, Alaska
  - Research Site, Tucson, Arizona
  - Research Site, Fayetteville, Arkansas
  - Research Site, Hot Springs, Arkansas
  - Research Site, Jonesboro, Arkansas
  - Research Site, Little Rock, Arkansas
  - Research Site, Anaheim, California
  - Research Site, Arcadia, California
  - Research Site, Berkeley, California
  - Research Site, Burbank, California
  - Research Site, Downey, California
  - Research Site, Fountain Valley, California
  - Research Site, Fresno, California
  - Research Site, La Verne, California
  - Research Site, Lancaster, California
  - Research Site, Long Beach, California
  - Research Site, Los Angeles, California
  - Research Site, Merced, California
  - Research Site, Mission Hills, California
  - Research Site, Montebello, California
  - Research Site, Oxnard, California
  - Research Site, Palm Springs, California
  - Research Site, Pismo Beach, California
  - Research Site, Pomona, California
  - Research Site, Redlands, California
  - Research Site, Salinas, California
  - Research Site, San Diego, California
  - Research Site, Santa Rosa, California
  - Research Site, Simi Valley, California
  - Research Site, Soquel, California
  - Research Site, St. Helena, California
  - Research Site, Torrance, California
  - Research Site, Vallejo, California
  - Research Site, West Covina, California
  - Research Site, Denver, Colorado
  - Research Site, Englewood, Colorado
  - Research Site, Bridgeport, Connecticut
  - Research Site, Southington, Connecticut
  - Research Site, Washington D.C., District of Columbia
  - Research Site, Boynton Beach, Florida
  - Research Site, Coral Springs, Florida
  - Research Site, Daytona Beach, Florida
  - Research Site, Fort Lauderdale, Florida
  - Research Site, Holiday, Florida
  - Research Site, Hollywood, Florida
  - Research Site, Jacksonville, Florida
  - Research Site, Kissimmee, Florida
  - Research Site, Lake Worth, Florida
  - Research Site, Lakeland, Florida
  - Research Site, Lecanto, Florida
  - Research Site, Miami, Florida
  - Research Site, New Port Richey, Florida
  - Research Site, Orange City, Florida
  - Research Site, Orlando, Florida
  - Research Site, Pembroke Pines, Florida
  - Research Site, Rockledge, Florida
  - Research Site, Tamarac, Florida
  - Research Site, The Villages, Florida
  - Research Site, Titusville, Florida
  - Research Site, Weston, Florida
  - Research Site, Albany, Georgia
  - Research Site, Augusta, Georgia
  - Research Site, Stockbridge, Georgia
  - Research Site, Thomasville, Georgia
  - Research Site, Chicago, Illinois
  - Research Site, Galesburg, Illinois
  - Research Site, Gurnee, Illinois
  - Research Site, Mount Vernon, Illinois
  - Research Site, Skokie, Illinois
  - Research Site, Indianapolis, Indiana
  - Research Site, Michigan City, Indiana
  - Research Site, Muncie, Indiana
  - Research Site, Council Bluffs, Iowa
  - Research Site, Dubuque, Iowa
  - Research Site, Iowa City, Iowa
  - Research Site, Sioux City, Iowa
  - Research Site, Waterloo, Iowa
  - Research Site, Hutchinson, Kansas
  - Research Site, Wichita, Kansas
  - Research Site, Ashland, Kentucky
  - Research Site, Hazard, Kentucky
  - Research Site, Louisville, Kentucky
  - Research Site, Morehead, Kentucky
  - Research Site, Mount Sterling, Kentucky
  - Research Site, Paducah, Kentucky
  - Research Site, Alexandria, Louisiana
  - Research Site, Lafayette, Louisiana
  - Research Site, Marrero, Louisiana
  - Research Site, New Orleans, Louisiana
  - Research Site, Ruston, Louisiana
  - Research Site, Shreveport, Louisiana
  - Research Site, Lewiston, Maine
  - Research Site, Rockport, Maine
  - Research Site, Baltimore, Maryland
  - Research Site, Bethesda, Maryland
  - Research Site, Chevy Chase, Maryland
  - Research Site, Cumberland, Maryland
  - Research Site, Frederick, Maryland
  - Research Site, Hagerstown, Maryland
  - Research Site, Towson, Maryland
  - Research Site, Westminster, Maryland
  - Research Site, Attleboro, Massachusetts
  - Research Site, Boston, Massachusetts
  - Research Site, Brockton, Massachusetts
  - Research Site, Cambridge, Massachusetts
  - Research Site, Worcester, Massachusetts
  - Research Site, Clarkston, Michigan
  - Research Site, Grand Rapids, Michigan
  - Research Site, Kalamazoo, Michigan
  - Research Site, Southfield, Michigan
  - Research Site, Southgate, Michigan
  - Research Site, Willmar, Minnesota
  - Research Site, Biloxi, Mississippi
  - Research Site, Hattiesburg, Mississippi
  - Research Site, Jackson, Mississippi
  - Research Site, Tupelo, Mississippi
  - Research Site, Columbia, Missouri
  - Research Site, Jefferson City, Missouri
  - Research Site, Kansas City, Missouri
  - Research Site, Springfield, Missouri
  - Research Site, St Louis, Missouri
  - Research Site, Great Falls, Montana
  - Research Site, Kalispell, Montana
  - Research Site, Grand Island, Nebraska
  - Research Site, Omaha, Nebraska
  - Research Site, Henderson, Nevada
  - Research Site, North Las Vegas, Nevada
  - Research Site, Manchester, New Hampshire
  - Research Site, Sparta, New Jersey
  - Research Site, Teaneck, New Jersey
  - Research Site, Vineland, New Jersey
  - Research Site, Albuquerque, New Mexico
  - Research Site, Santa Fe, New Mexico
  - Research Site, Albany, New York
  - Research Site, Brooklyn, New York
  - Research Site, Buffalo, New York
  - Research Site, Glens Falls, New York
  - Research Site, Goshen, New York
  - Research Site, Lake Success, New York
  - Research Site, Latham, New York
  - Research Site, Nyack, New York
  - Research Site, Poughkeepsie, New York
  - Research Site, Staten Island, New York
  - Research Site, Syracuse, New York
  - Research Site, Valhalla, New York
  - Research Site, Asheboro, North Carolina
  - Research Site, Asheville, North Carolina
  - Research Site, Burlington, North Carolina
  - Research Site, Concord, North Carolina
  - Research Site, Durham, North Carolina
  - Research Site, Goldsboro, North Carolina
  - Research Site, Greenville, North Carolina
  - Research Site, Hendersonville, North Carolina
  - Research Site, Hickory, North Carolina
  - Research Site, High Point, North Carolina
  - Research Site, Huntersville, North Carolina
  - Research Site, Kinston, North Carolina
  - Research Site, Pinehurst, North Carolina
  - Research Site, Raleigh, North Carolina
  - Research Site, Washington, North Carolina
  - Research Site, Bismarck, North Dakota
  - Research Site, Akron, Ohio
  - Research Site, Columbus, Ohio
  - Research Site, Dayton, Ohio
  - Research Site, Massillon, Ohio
  - Research Site, Middletown, Ohio
  - Research Site, Port Clinton, Ohio
  - Research Site, Sylvania, Ohio
  - Research Site, Wooster, Ohio
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, Tulsa, Oklahoma
  - Research Site, Bethlehem, Pennsylvania
  - Research Site, Gettysburg, Pennsylvania
  - Research Site, Langhorne, Pennsylvania
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Pittsburgh, Pennsylvania
  - Research Site, Upland, Pennsylvania
  - Research Site, Willow Grove, Pennsylvania
  - Research Site, Wynnewood, Pennsylvania
  - Research Site, Pawtucket, Rhode Island
  - Research Site, Providence, Rhode Island
  - Research Site, Woonsocket, Rhode Island
  - Research Site, Aiken, South Carolina
  - Research Site, Charleston, South Carolina
  - Research Site, Columbia, South Carolina
  - Research Site, Hilton Head Island, South Carolina
  - Research Site, Myrtle Beach, South Carolina
  - Research Site, Sumter, South Carolina
  - Research Site, Aberdeen, South Dakota
  - Research Site, Sioux Falls, South Dakota
  - Research Site, Watertown, South Dakota
  - Research Site, Johnson City, Tennessee
  - Research Site, Knoxville, Tennessee
  - Research Site, Memphis, Tennessee
  - Research Site, Nashville, Tennessee
  - Research Site, Abilene, Texas
  - Research Site, Amarillo, Texas
  - Research Site, Austin, Texas
  - Research Site, Beaumont, Texas
  - Research Site, Bedford, Texas
  - Research Site, Bryan, Texas
  - Research Site, Corpus Christi, Texas
  - Research Site, Dallas, Texas
  - Research Site, El Paso, Texas
  - Research Site, Fort Worth, Texas
  - Research Site, Garland, Texas
  - Research Site, Harlingen, Texas
  - Research Site, Houston, Texas
  - Research Site, Irving, Texas
  - Research Site, Longview, Texas
  - Research Site, McAllen, Texas
  - Research Site, Mesquite, Texas
  - Research Site, Midland, Texas
  - Research Site, Paris, Texas
  - Research Site, Richardson, Texas
  - Research Site, Round Rock, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Sherman, Texas
  - Research Site, Southlake, Texas
  - Research Site, Sugar Land, Texas
  - Research Site, Temple, Texas
  - Research Site, The Woodlands, Texas
  - Research Site, Tyler, Texas
  - Research Site, Waco, Texas
  - Research Site, Webster, Texas
  - Research Site, Wichita Falls, Texas
  - Research Site, Ogden, Utah
  - Research Site, White River Junction, Vermont
  - Research Site, Christiansburg, Virginia
  - Research Site, Fairfax, Virginia
  - Research Site, Lynchburg, Virginia
  - Research Site, Newport News, Virginia
  - Research Site, Portsmouth, Virginia
  - Research Site, Bremerton, Washington
  - Research Site, Burien, Washington
  - Research Site, Edmonds, Washington
  - Research Site, Seattle, Washington
  - Research Site, Spokane, Washington
  - Research Site, Tacoma, Washington
  - Research Site, Vancouver, Washington
  - Research Site, Yakima, Washington
  - Research Site, Green Bay, Wisconsin
  - Research Site, Janesville, Wisconsin
  - Research Site, Milwaukee, Wisconsin
- Argentina (9):
  - Research Site, Quilmes, Buenos Aires
  - Research Site, Córdoba, Córdoba Province
  - Research Site, Buenos Aires, Distrito Federal
  - Research Site, San Salvador de Jujuy, Jujuy Province
  - Research Site, Rosario, Santa Fe Province
  - Research Site, San Miguel de Tucumán, Tucumán Province
  - Research Site, Buenos Aires
  - Research Site, La Rioja
  - Research Site, Santa Fe
- Austria (2):
  - Research Site, Steyr
  - Research Site, Vienna
- Belgium (5):
  - Research Site, Ieper
  - Research Site, Libramont
  - Research Site, Liège
  - Research Site, Namur
  - Research Site, Ottignies
- Brazil (21):
  - Research Site, Fortaleza, Ceará
  - Research Site, Cachoeiro de Itapemirim, Espírito Santo
  - Research Site, Salvador, Estado de Bahia
  - Research Site, Brasília, Federal District
  - Research Site, Campo Grande, Mato Grosso do Sul
  - Research Site, Belo Horizonte, Minas Gerais
  - Research Site, Curitba, Paraná
  - Research Site, Curitiba, Paraná
  - Research Site, Londrina, Paraná
  - Research Site, Belém, Pará
  - Research Site, Ijuí, Rio Grande do Sul
  - Research Site, Passo Fundo, Rio Grande do Sul
  - Research Site, Pelotas, Rio Grande do Sul
  - Research Site, Porto Alegre, Rio Grande do Sul
  - Research Site, Itajaí, Santa Catarina
  - Research Site, Ribeirão Preto, São Paulo
  - Research Site, Santo André, São Paulo
  - Research Site, São José dos Campos, São Paulo
  - Research Site, São Paulo, São Paulo
  - Research Site, Rio de Janeiro
  - Research Site, São Paulo
- Bulgaria (3):
  - Research Site, Rousse
  - Research Site, Sofia
  - Research Site, Varna
- Canada (5):
  - Research Site, Moncton, New Brunswick
  - Research Site, Oshawa, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Montreal, Quebec
  - Research Site, Saint-Jérôme, Quebec
- Chile (3):
  - Research Site, Temuco, Cautín
  - Research Site, Reñaca, Región de Valparaíso
  - Research Site, Santiago
- China (26):
  - Research Site, Beijing, Beijing Municipality
  - Research Site, Chongqing, Chongqing Municipality
  - Research Site, Fuzhou, Fujian
  - Research Site, Lanzhou, Gansu
  - Research Site, Guangzhou, Guangdong
  - Research Site, Zhongshan, Guangdong
  - Research Site, Haikou, Hainan
  - Research Site, Shijiazhuang, Hebei
  - Research Site, Harbin, Heilongjiang
  - Research Site, Wuhan, Hubei
  - Research Site, Changsha, Hunan
  - Research Site, Nanjing, Jiangsu
  - Research Site, Suzhou, Jiangsu
  - Research Site, Nanchang, Jiangxi
  - Research Site, Changchun, Jilin
  - Research Site, Dalian, Liaoning
  - Research Site, Shenyang, Liaoning
  - Research Site, Xi'an, Shaanxi
  - Research Site, Jinan, Shandong
  - Research Site, Chengdu, Sichuan
  - Research Site, Ürümqi, Xinjiang
  - Research Site, Kunming, Yunnan
  - Research Site, Hangzhou, Zhejiang
  - Research Site, Beijing
  - Research Site, Chongqing
  - Research Site, Shanghai
- Croatia (2):
  - Research Site, Rijeka
  - Research Site, Zagreb
- Czechia (8):
  - Research Site, Benesov U Prahy
  - Research Site, Hořovice
  - Research Site, Kutná Hora
  - Research Site, Kyjov
  - Research Site, Nová Ves pod Pleší
  - Research Site, Ostrava-Poruba
  - Research Site, Prague
  - Research Site, Příbram
- Germany (5):
  - Research Site, Bad Berka
  - Research Site, Köln-Merheim
  - Research Site, Moers
  - Research Site, München
  - Research Site, Münster
- Greece (6):
  - Research Site, Athens
  - Research Site, Chania
  - Research Site, Larissa
  - Research Site, Nea Kifissia, Athens
  - Research Site, Piraeus
  - Research Site, Thessaloniki
- Hong Kong (3):
  - Research Site, Hong Kong
  - Research Site, Kowloon
  - Research Site, New Territories
- India (15):
  - Research Site, Panjim, Goa
  - Research Site, Ahmedabad, Gujarat
  - Research Site, Bangalore, Karnataka
  - Research Site, Mangalore, Karnataka
  - Research Site, Kochi, Kerala
  - Research Site, Bhopal, Madhya Pradesh
  - Research Site, Ahilyanagar, Maharashtra
  - Research Site, Aurangabad, Maharashtra
  - Research Site, Thane, Maharashtra
  - Research Site, New Delhi, National Capital Territory of Delhi
  - Research Site, Jaipur, Rajasthan
  - Research Site, Chennai, Tamil Nadu
  - Research Site, Madurai, Tamil Nadu
  - Research Site, Kolkata, West Bengal
  - Research Site, Bangalore
- Research Site, Dublin, Ireland
- Israel (5):
  - Research Site, Jerusalem
  - Research Site, Kfar Saba
  - Research Site, Poria Eylit
  - Research Site, Rehovot
  - Research Site, Tel Aviv
- Italy (13):
  - Research Site, Catania
  - Research Site, Faenza RA
  - Research Site, Grosseto
  - Research Site, Lecce
  - Research Site, Legnago VR
  - Research Site, Lugo RA
  - Research Site, Meldola FC
  - Research Site, Messina
  - Research Site, Milan
  - Research Site, Napoli
  - Research Site, Ravenna
  - Research Site, Reggio Calabria
  - Research Site, San Giovanni Rotondo FG
- Japan (15):
  - Research Site, Nagoya, Aichi-ken
  - Research Site, Fukui-shi, Fukui
  - Research Site, Chikushino-shi, Fukuoka
  - Research Site, Kurume-shi, Fukuoka
  - Research Site, Amagasaki-shi, Hyōgo
  - Research Site, Kobe, Hyōgo
  - Research Site, Nishinomiya-shi, Hyōgo
  - Research Site, Kanazawa, Ishikawa-ken
  - Research Site, Sagamihara-shi, Kanagawa
  - Research Site, Okayama, Okayama-ken
  - Research Site, Osaka, Osaka
  - Research Site, Bunkyo-ku, Tokyo
  - Research Site, Shinjuku-ku, Tokyo
  - Research Site, Yonago-shi, Tottori
  - Research Site, Kyoto
- Luxembourg (2):
  - Research Site, Esch-sur-Alzette
  - Research Site, Luxembourg
- Malaysia (5):
  - Research Site, Kota Bharu, Kelantan
  - Research Site, Kuala Lumpur, Kuala Lumpur
  - Research Site, Kuantan, Pahang
  - Research Site, George Town, Pulau Pinang
  - Research Site, Kota Kinabalu, Sabah
- Mexico (13):
  - Research Site, Saltillo, Coahuila
  - Research Site, León, Guanajuato
  - Research Site, Guadalajara, Jalisco
  - Research Site, Zapopan, Jalisco
  - Research Site, Mexico City, Mexico City
  - Research Site, Monterrey, Nuevo León
  - Research Site, Querétaro City, Querétaro
  - Research Site, San Luis Potosí City, San Luis Potosí
  - Research Site, Mérida, Yucatán
  - Research Site, Chihuahua City
  - Research Site, Colima
  - Research Site, Oaxaca City
  - Research Site, Puebla City
- Netherlands (4):
  - Research Site, Breda
  - Research Site, Eindhoven
  - Research Site, Rotterdam
  - Research Site, Tilburg
- Research Site, Davao City, Davao Region, Philippines
- Poland (3):
  - Research Site, Krakow
  - Research Site, Olsztyn
  - Research Site, Rzeszów
- Research Site, San Juan, Puerto Rico
- Research Site, Sibiu, Romania
- Russia (26):
  - Research Site, Arkhangelsk
  - Research Site, Barnaul
  - Research Site, Belgorod
  - Research Site, Ivanovo
  - Research Site, Kirov
  - Research Site, Krasnodar
  - Research Site, Kursk
  - Research Site, Lipetsk
  - Research Site, Moscow
  - Research Site, Nizhny Novgorod
  - Research Site, Novosibirsk
  - Research Site, Obninsk
  - Research Site, Omsk
  - Research Site, Orenburg
  - Research Site, Penza
  - Research Site, Pyatigorsk
  - Research Site, Saint Petersburg
  - Research Site, Samara
  - Research Site, Saratov
  - Research Site, Stavropol
  - Research Site, Tula
  - Research Site, Tver'
  - Research Site, Ufa
  - Research Site, Ulyanovsk
  - Research Site, Voronezh
  - Research Site, Yaroslavl
- Serbia (4):
  - Research Site, Belgrade
  - Research Site, Gornji Matejevac
  - Research Site, Kamenitz
  - Research Site, Kragujevac
- Slovenia (2):
  - Research Site, Golnik
  - Research Site, Pohorje
- South Africa (5):
  - Research Site, Umhlanga, KwaZulu-Natal
  - Research Site, Bloemfontein
  - Research Site, Johannesburg
  - Research Site, Overport
  - Research Site, Polokwane
- South Korea (3):
  - Research Site, Gwangju
  - Research Site, Seongnam-si, Gyeonggido
  - Research Site, Seoul
- Spain (7):
  - Research Site, Granada, Andalusia
  - Research Site, Las Palmas de Gran Canaria, Canary Islands
  - Research Site, Barcelona, Catalonia
  - Research Site, Pontevedra, Galicia
  - Research Site, Alicante, Valencia
  - Research Site, Benidorm, Valencia
  - Research Site, Valencia, Valencia
- Switzerland (4):
  - Research Site, Aarau
  - Research Site, Chur
  - Research Site, Sursee
  - Research Site, Zurich
- Taiwan (2):
  - Research Site, Kaohsiung City
  - Research Site, Taichung
- Research Site, Kirovograd, Ukraine
- United Kingdom (5):
  - Research Site, Bebington
  - Research Site, Dorechester
  - Research Site, Dorset
  - Research Site, Liverpool
  - Research Site, Manchester

REFERENCES:
- [Background] Gascon P, Nagarkar R, Smakal M, Syrigos KN, Barrios CH, Sanchez JC, Zhang L, Henry DH, Gordon D, Hirsh V, Kubota K, Orlov S, Thomas G, Steinmetz T, Kang JH, Tomita DK, Fleishman AN, Park JK, De Oliveira Brandao C. A Randomized, Double-Blind, Placebo-Controlled, Phase III Noninferiority Study of the Long-Term Safety and Efficacy of Darbepoetin Alfa for Chemotherapy-Induced Anemia in Patients With Advanced NSCLC. J Thorac Oncol. 2020 Feb;15(2):190-202. doi: 10.1016/j.jtho.2019.10.005. Epub 2019 Oct 16. PMID 31629060
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 371 centers in Europe, Latin America, Asia, India, North America, Israel, and South Africa.
Pre-assignment Details: Eligible participants were randomized to darbepoetin alfa or placebo in a 2:1 ratio. Randomization was stratified by histology (squamous vs other), screening hemoglobin (< 10.0 g/dL vs ≥ 10.0 g/dL), and geographic region.
Period: Overall Study
Arm/Group | Placebo | Darbepoetin Alfa
Started | 846 | 1703
Received Study Drug | 837 | 1681
Completed (Participants who died) | 642 | 1246
Not Completed | 204 | 457
Not completed — Administrative Decision | 3 | 2
Not completed — Adverse Event | 5 | 2
Not completed — Withdrawal by Subject | 44 | 118
Not completed — Ineligibility Determined | 1 | 10
Not completed — Lost to Follow-up | 24 | 54
Not completed — Noncompliance | 3 | 4
Not completed — Protocol Deviation | 0 | 2
Not completed — Other | 9 | 17
Not completed — Missing | 1 | 1
Not completed — Still on-study | 114 | 247

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Darbepoetin Alfa | Total
Number analyzed (Participants) | 846 | 1703 | 2549
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.2 (9.9) | 61.6 (9.8) | 61.8 (9.8)
Age, Customized [Count of Participants; unit: Participants]
  18 - 64 years | 482 | 1014 | 1496
  65 - 74 years | 287 | 547 | 834
  75 - 84 years | 71 | 134 | 205
  ≥ 85 years | 6 | 8 | 14
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 281 | 585 | 866
  Male | 565 | 1118 | 1683
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White or Caucasian | 404 | 808 | 1212
  Black or African American | 27 | 46 | 73
  Asian | 357 | 741 | 1098
  Japanese | 7 | 12 | 19
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Aborigine | 0 | 1 | 1
  Other | 5 | 14 | 19
  Hispanic | 45 | 81 | 126
Geographic Region [Count of Participants; unit: Participants] — Stratification factor at the time of randomization. Population: The primary analysis set includes all randomized and consented participants with non-small cell lung cancer who received at least one dose of study drug.
  Participants
    number analyzed (Participants) | 836 | 1680 | 2516
    Western Europe, Israel and South Africa | 54 | 108 | 162
    Central and Eastern Europe | 220 | 451 | 671
    Latin America and Asia | 166 | 337 | 503
    India | 168 | 339 | 507
    North America | 99 | 192 | 291
    China | 123 | 243 | 366
    Japan | 6 | 10 | 16
Histology [Count of Participants; unit: Participants] — Stratification factor at the time of randomization Population: Primary analysis set
  Participants
    number analyzed (Participants) | 836 | 1680 | 2516
    Squamous | 289 | 589 | 878
    Non-squamous | 547 | 1091 | 1638
Screening Hemoglobin [Count of Participants; unit: Participants] — Stratification factor at the time of randomization. Population: Primary analysis set
  Participants
    number analyzed (Participants) | 836 | 1680 | 2516
    < 10 g/dL | 433 | 870 | 1303
    ≥ 10 g/dL | 403 | 810 | 1213

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS)
Description: Overall survival (OS) was defined as the time from randomization to the date of death due to any cause. Participants were censored on the date of last contact (ie, the date the participant was last known to be alive) if they were not known to have died.
Time Frame: From randomization until death or end of study; maximum time on follow-up was 93.6 months.
Population: Primary analysis set (all randomized and consented participants with non-small cell lung cancer who received at least one dose of study drug)
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Placebo | Darbepoetin Alfa
Number analyzed (Participants) | 836 | 1680
months | 9.260 [8.250 to 10.020] | 9.460 [8.900 to 10.120]
Statistical Analysis 1: Comparison: Placebo vs Darbepoetin Alfa; The primary analysis used the Cox Proportional Hazard Model stratified by the randomization stratification factors (geographic region, histology, and screening hemoglobin), with treatment group as the only covariate; Test type: Non-Inferiority — Non-inferiority was declared if the upper confidence limit for the hazard ratio (darbepoetin alfa to placebo) was less than 1.15 using a 1-sided significance level of 0.025; Hazard Ratio (HR) = 0.92, 95% CI 2-sided [0.83 to 1.01] — A hazard ratio < 1.0 indicates a lower risk of death for darbepoetin alfa relative to placebo
Statistical Analysis 2: Comparison: Placebo vs Darbepoetin Alfa; As a sensitivity analysis, an unstratified Cox Proportional Hazard Model with treatment group as the only covariate was conducted; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.91, 95% CI 2-sided [0.83 to 1.00] — A hazard ratio < 1.0 indicates a lower risk of death for darbepoetin alfa relative to placebo
Statistical Analysis 3: Comparison: Placebo vs Darbepoetin Alfa; Test type: Superiority — If non-inferiority was demonstrated for both OS and PFS and superiority was demonstrated for the transfusion endpoint, superiority was then tested for both OS and PFS using the Hochberg procedure to adjust for multiplicity; p = 0.070, Stratified log-rank test; Stratified by the randomization stratification factors (geographic region, histology, screening hemoglobin)
Statistical Analysis 4: Comparison: Placebo vs Darbepoetin Alfa; Test type: Superiority; p = 0.047, Log Rank; Unstratified log rank test
Statistical Analysis 5: Comparison: Placebo vs Darbepoetin Alfa; To evaluate the potential effect of cross-in (participants in the placebo group who began treatment with an erythropoiesis-stimulating agent (ESA) at any point after randomization), a sensitivity analysis was conducted that included ESA use as a time-dependent covariate in a Cox regression model stratified by the randomization stratification factors (geographic region, histology, and screening hemoglobin); Test type: Other; Hazard Ratio (HR) = 0.93, 95% CI 2-sided [0.84 to 1.02]

2. Secondary Outcome: Progression-free Survival (PFS)
Description: Progression-free survival was defined as the time from randomization to the date of radiographic disease progression or death from any cause, whichever event occurred first. Participants without either event were censored on the date of their last disease assessment. Disease progression was based on the investigator's assessment of scans using the Response Evaluation Criteria in Solid Tumors (RECIST) version 1.0 or 1.1 depending on the timing of enrollment.
Time Frame: From randomization until disease progression or death; maximum time on follow-up was 87.23 months.
Population: The radiographic endpoint primary analysis set includes all participants in the primary analysis set who did not have disease progression prior to randomization.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Placebo | Darbepoetin Alfa
Number analyzed (Participants) | 819 | 1638
months | 4.340 [4.170 to 4.700] | 4.800 [4.370 to 5.320]
Statistical Analysis 1: Comparison: Placebo vs Darbepoetin Alfa; The primary analysis of PFS used a Cox Proportional Hazard Model stratified by the randomization stratification factors (geographic region, histology, and screening hemoglobin), with treatment group as the only covariate; Test type: Non-Inferiority — If non-inferiority was declared for OS, non-inferiority would be declared for PFS if the upper confidence limit for the hazard ratio was less than 1.15 using a 1-sided significance level of 0.025; Hazard Ratio (HR) = 0.95, 95% CI 2-sided [0.87 to 1.04] — A hazard ratio < 1.0 indicates a lower risk of death or progression for darbepoetin alfa relative to placebo
Statistical Analysis 2: Comparison: Placebo vs Darbepoetin Alfa; [analysis description as in outcome 1, analysis 2]; Test type: Non-Inferiority — [test comment as in outcome 2, analysis 1]; Hazard Ratio (HR) = 0.95, 95% CI 2-sided [0.87 to 1.04] — A hazard ratio < 1.0 indicates a lower risk of death or progression for darbepoetin alfa relative to placebo
Statistical Analysis 3: Comparison: Placebo vs Darbepoetin Alfa; Test type: Superiority — [test comment as in outcome 1, analysis 3]; p = 0.31, Stratified log-rank test; Stratified by the randomization stratification factors (geographic region, histology, screening hemoglobin)
Statistical Analysis 4: Comparison: Placebo vs Darbepoetin Alfa; Test type: Superiority; p = 0.27, Log Rank; Unstratified log rank test
Statistical Analysis 5: Comparison: Placebo vs Darbepoetin Alfa; [analysis description as in outcome 1, analysis 5]; Test type: Other; Hazard Ratio (HR) = 0.96, 95% CI 2-sided [0.88 to 1.05]

3. Secondary Outcome: Percentage of Participants With a Red Blood Cell Transfusion or Hemoglobin ≤ 8.0 g/dL From Week 5 to End of the Efficacy Treatment Period
Description: Any red blood cell (RBC) transfusion (packed RBCs or whole blood) given or a hemoglobin ≤ 8.0 g/dL on or after study day 29 until the EOETP, inclusive.
Time Frame: Week 5 (day 29) to end of the efficacy treatment period (EOETP; defined as 21 days after either the last dose of study drug or the last dose of chemotherapy, whichever was later); median (range) duration of dosing was 10 (1 to 106) weeks in both groups.
Population: Primary analysis set participants who were on study as of day 29
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Darbepoetin Alfa
Number analyzed (Participants) | 764 | 1517
percentage of participants | 29.2 | 22.5
Statistical Analysis 1: Comparison: Placebo vs Darbepoetin Alfa; The primary analysis of the incidence of a transfusion or hemoglobin ≤ 8.0 g/dL from day 29 to EOETP was based on the Cochran-Mantel-Haenszel method to test for treatment group differences while adjusting for the randomization stratification factors (geographic region, histology, and screening hemoglobin); Test type: Superiority — If non-inferiority was declared for OS and PFS, superiority would be declared for the transfusion endpoint if the p-value from a two-sided test of significance using the Cochran-Mantel-Haenszel method was less than 0.05 in favor of the darbepoetin alfa group; p < 0.001, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.704, 95% CI 2-sided [0.573 to 0.864] — An odds ratio < 1.0 indicates a lower event rate for darbepoetin alfa relative to placebo
Statistical Analysis 2: Comparison: Placebo; As a sensitivity analysis a logistic regression analysis was conducted, stratified by the randomization stratification factors (geographic region, histology, screening hemoglobin); Test type: Other; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 0.705, 95% CI 2-sided [0.574 to 0.866] — An odds ratio < 1.0 indicates a lower event rate for darbepoetin alfa relative to placebo

4. Secondary Outcome: Number of Participants With Adverse Events of Special Interest
Description: Adverse events of interest for darbepoetin alfa, based on clinical data in anemic patients with cancer to date, included the following categories: antibody-mediated pure red cell aplasia (PRCA), cardiac failure, central nervous system vascular disorders, convulsions, embolic and thrombotic events, hypersensitivity, hypertension, ischemic heart disease, malignancies, and severe cutaneous adverse reactions. Lack of efficacy and medication errors were also evaluated.
Time Frame: From first dose of study drug until 30 days after last dose; the median (range) duration of treatment was 10 (1 to 106) weeks in both groups.
Population: All randomized and consented participants who received at least 1 dose of study drug. Four participants in the placebo group received at least 1 dose of darbepoetin alfa during the study and were included in the darbepoetin alfa group for safety analyses.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Darbepoetin Alfa
Number analyzed (Participants) | 833 | 1685
Participants
  Any adverse events of interest | 157 | 369
  Antibody-mediated pure red cell aplasia | 20 | 51
  Cardiac failure | 7 | 12
  Central nervous system vascular disorders | 8 | 25
  Convulsions | 8 | 9
  Embolic and thrombotic events | 34 | 89
  Embolic and thrombotic events, arterial | 6 | 19
  Embolic and thrombotic events, venous | 23 | 51
  Embolic and thrombotic events, unspecified/mixed | 10 | 26
  Hypersensitivity | 75 | 178
  Hypertension | 26 | 41
  Ischaemic heart disease | 9 | 23
  Lack of efficacy/effect | 0 | 0
  Malignancies | 16 | 38
  Medication errors | 0 | 1
  Severe cutaneous adverse reactions | 11 | 35

5. Secondary Outcome: Percentage of Participants With an Objective Tumor Response
Description: Objective response was defined as the incidence of a complete or partial response at any time during the study. Response was determined by the investigator's assessment of the scans using RECIST version 1.0 or 1.1 depending on the timing of enrollment.
Time Frame: Day 1 to end of the efficacy treatment period (EOETP; defined as 21 days after either the last dose of study drug or the last dose of chemotherapy, whichever was later); median (range) duration of dosing was 10 (1 to 106) weeks in both groups.
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Darbepoetin Alfa
Number analyzed (Participants) | 819 | 1638
percentage of participants | 32.6 | 36.2
Statistical Analysis 1: Comparison: Placebo vs Darbepoetin Alfa; Test type: Other; p = 0.076, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel method adjusted for the randomization stratification factors (geographic region, histology, screening hemoglobin); Odds Ratio (OR) = 1.173, 95% CI 2-sided [0.983 to 1.401] — An odds ratio < 1.0 indicates a lower event rate for darbepoetin alfa relative to placebo
Statistical Analysis 2: Comparison: Placebo vs Darbepoetin Alfa; Test type: Other; p = 0.078, Cochran-Mantel-Haenszel; Unstratified analysis; Odds Ratio (OR) = 1.173, 95% CI 2-sided [0.982 to 1.401]

6. Secondary Outcome: Number of Participants Who Developed Neutralizing Antibodies to Darbepoetin Alfa
Description: Developing antibody incidence was defined as neutralizing antibody positive postbaseline with a negative or no result at baseline.
Time Frame: Baseline and end of the efficacy treatment period (EOETP; defined as 21 days after either the last dose of study drug or the last dose of chemotherapy, whichever was later. the median (range) duration of treatment was 10 (1 to 106) weeks in both groups.
Population: Randomized and consented participants who received at least one dose of study drug and with a postbaseline result.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Darbepoetin Alfa
Number analyzed (Participants) | 803 | 1606
Participants | 0 | 0

7. Secondary Outcome: Percentage of Participants With a Red Blood Cell Transfusion or Hemoglobin ≤ 8.0 g/dL From Week 1 to End of the Efficacy Treatment Period
Description: Any red blood cell (RBC) transfusion (packed RBCs or whole blood) given or a hemoglobin ≤ 8.0 g/dL on or after study day 1 until the EOETP, inclusive.
Time Frame: Week 1 to end of the efficacy treatment period (EOETP; defined as 21 days after either the last dose of study drug or the last dose of chemotherapy, whichever was later); the median (range) duration of treatment was 10 (1 to 106) weeks in both groups.
Population: Primary analysis set
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Darbepoetin Alfa
Number analyzed (Participants) | 836 | 1680
percentage of participants | 29.7 | 24.2
Statistical Analysis 1: Comparison: Placebo vs Darbepoetin Alfa; Test type: Other; p = 0.003, Cochran-Mantel-Haenszel; [statistical method as in outcome 5, analysis 1]; Odds Ratio (OR) = 0.741, 95% CI 2-sided [0.610 to 0.901] — An odds ratio < 1.0 indicates a lower event rate for darbepoetin alfa relative to placebo
Statistical Analysis 2: Comparison: Placebo vs Darbepoetin Alfa; Test type: Other; p = 0.003, Cochran-Mantel-Haenszel; Unstratified analysis; Odds Ratio (OR) = 0.758, 95% CI 2-sided [0.630 to 0.913]

8. Secondary Outcome: Change From Baseline in Hemoglobin to End of Efficacy Treatment Period
Description: Post-baseline hemoglobin values within 28 days after a RBC transfusion were not be used in the calculation of change.
Time Frame: Baseline and end of the efficacy treatment period (EOETP; defined as 21 days after either the last dose of study drug or the last dose of chemotherapy, whichever was later); the median (range) duration of treatment was 10 (1 to 106) weeks in both groups.
Population: Primary analysis set with available baseline and at least 1 postbaseline value; if the EOETP value was missing, the last available postbaseline value was used.
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Placebo | Darbepoetin Alfa
Number analyzed (Participants) | 633 | 1344
g/dL | -0.11 (1.71) | 0.50 (1.81)

ADVERSE EVENTS:
Time Frame: From first dose of study drug until 30 days after last dose; the median (range) duration of treatment was 10 (1 to 106) weeks in both groups.
Description: The safety population included all randomized and consented participants who received at least 1 dose of study drug. Four participants in the placebo group received at least 1 dose of darbepoetin alfa during the study and were included in the darbepoetin alfa group for safety analyses.
  Other Adverse Events summarizes the non-serious occurrences of adverse events that exceed the indicated frequency threshold.
Arm/Group | Placebo | Darbepoetin Alfa
All-Cause Mortality (participants affected / at risk) | 657/833 | 1273/1685
Serious Adverse Events (participants affected / at risk) | 259/833 | 524/1685
Other Adverse Events (participants affected / at risk) | 674/833 | 1319/1685
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=833) | Darbepoetin Alfa (N=1685)
Anaemia (Blood and lymphatic system disorders) | 46 | 57
Bicytopenia (Blood and lymphatic system disorders) | 0 | 1
Bone marrow failure (Blood and lymphatic system disorders) | 8 | 20
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 7 | 14
Haemolytic anaemia (Blood and lymphatic system disorders) | 0 | 1
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 1 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 1
Leukopenia (Blood and lymphatic system disorders) | 2 | 7
Neutropenia (Blood and lymphatic system disorders) | 6 | 17
Pancytopenia (Blood and lymphatic system disorders) | 4 | 9
Sideroblastic anaemia (Blood and lymphatic system disorders) | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 16 | 28
Thrombocytosis (Blood and lymphatic system disorders) | 0 | 1
Acute coronary syndrome (Cardiac disorders) | 1 | 3
Acute myocardial infarction (Cardiac disorders) | 3 | 5
Angina pectoris (Cardiac disorders) | 1 | 1
Arrhythmia (Cardiac disorders) | 0 | 2
Atrial fibrillation (Cardiac disorders) | 3 | 8
Atrioventricular block complete (Cardiac disorders) | 1 | 0
Cardiac arrest (Cardiac disorders) | 2 | 7
Cardiac failure (Cardiac disorders) | 0 | 1
Cardiac failure acute (Cardiac disorders) | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 2 | 1
Cardiac tamponade (Cardiac disorders) | 1 | 1
Cardio-respiratory arrest (Cardiac disorders) | 7 | 9
Cardio-respiratory distress (Cardiac disorders) | 1 | 1
Cardiogenic shock (Cardiac disorders) | 1 | 1
Cardiopulmonary failure (Cardiac disorders) | 2 | 2
Cardiovascular insufficiency (Cardiac disorders) | 1 | 0
Left ventricular dysfunction (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 1 | 5
Myocardial ischaemia (Cardiac disorders) | 0 | 2
Nodal arrhythmia (Cardiac disorders) | 0 | 1
Pericardial effusion (Cardiac disorders) | 1 | 2
Sinus node dysfunction (Cardiac disorders) | 0 | 1
Sinus tachycardia (Cardiac disorders) | 0 | 1
Ventricular fibrillation (Cardiac disorders) | 0 | 1
Vertigo (Ear and labyrinth disorders) | 1 | 1
Adrenal insufficiency (Endocrine disorders) | 0 | 1
Toxic nodular goitre (Endocrine disorders) | 0 | 1
Angle closure glaucoma (Eye disorders) | 0 | 1
Retinal detachment (Eye disorders) | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 2
Abdominal pain (Gastrointestinal disorders) | 0 | 12
Abdominal pain upper (Gastrointestinal disorders) | 0 | 2
Constipation (Gastrointestinal disorders) | 0 | 4
Diarrhoea (Gastrointestinal disorders) | 8 | 12
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 0 | 1
Dysphagia (Gastrointestinal disorders) | 1 | 1
Enterocolitis (Gastrointestinal disorders) | 0 | 1
Faecaloma (Gastrointestinal disorders) | 0 | 1
Faeces discoloured (Gastrointestinal disorders) | 0 | 1
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 2
Gastrointestinal motility disorder (Gastrointestinal disorders) | 0 | 1
Haematemesis (Gastrointestinal disorders) | 1 | 1
Ileus (Gastrointestinal disorders) | 1 | 0
Incarcerated inguinal hernia (Gastrointestinal disorders) | 1 | 0
Intestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Large intestine perforation (Gastrointestinal disorders) | 0 | 2
Melaena (Gastrointestinal disorders) | 1 | 1
Nausea (Gastrointestinal disorders) | 2 | 3
Necrotising colitis (Gastrointestinal disorders) | 0 | 1
Neutropenic colitis (Gastrointestinal disorders) | 0 | 1
Oesophageal ulcer (Gastrointestinal disorders) | 0 | 1
Peritoneal haemorrhage (Gastrointestinal disorders) | 1 | 0
Small intestinal perforation (Gastrointestinal disorders) | 0 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 2
Vomiting (Gastrointestinal disorders) | 2 | 9
Asthenia (General disorders) | 7 | 11
Chest pain (General disorders) | 2 | 5
Chills (General disorders) | 0 | 1
Death (General disorders) | 9 | 12
Disease progression (General disorders) | 1 | 1
Fatigue (General disorders) | 2 | 2
General physical health deterioration (General disorders) | 2 | 3
Inflammation (General disorders) | 0 | 1
Malaise (General disorders) | 1 | 2
Multiple organ dysfunction syndrome (General disorders) | 4 | 7
Non-cardiac chest pain (General disorders) | 0 | 5
Organ failure (General disorders) | 0 | 1
Pain (General disorders) | 1 | 4
Performance status decreased (General disorders) | 0 | 1
Pyrexia (General disorders) | 3 | 15
Sudden cardiac death (General disorders) | 1 | 2
Sudden death (General disorders) | 8 | 12
Swelling (General disorders) | 0 | 1
Systemic inflammatory response syndrome (General disorders) | 0 | 1
Cholangitis (Hepatobiliary disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 1
Hepatic failure (Hepatobiliary disorders) | 1 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 0
Anaphylactic reaction (Immune system disorders) | 1 | 0
Hypersensitivity (Immune system disorders) | 0 | 1
Transfusion associated graft versus host disease (Immune system disorders) | 0 | 1
Abdominal abscess (Infections and infestations) | 1 | 0
Abscess (Infections and infestations) | 1 | 0
Appendicitis (Infections and infestations) | 1 | 0
Bacteraemia (Infections and infestations) | 0 | 1
Bacterial sepsis (Infections and infestations) | 0 | 1
Bronchitis (Infections and infestations) | 3 | 2
Cellulitis (Infections and infestations) | 1 | 3
Clostridium difficile colitis (Infections and infestations) | 0 | 1
Cystitis (Infections and infestations) | 1 | 0
Dengue fever (Infections and infestations) | 0 | 1
Device related infection (Infections and infestations) | 1 | 1
Empyema (Infections and infestations) | 1 | 2
Endometritis (Infections and infestations) | 0 | 1
Erysipelas (Infections and infestations) | 1 | 0
Furuncle (Infections and infestations) | 0 | 1
Gangrene (Infections and infestations) | 2 | 2
Gastroenteritis (Infections and infestations) | 2 | 7
Gastroenteritis viral (Infections and infestations) | 0 | 1
Hepatitis B (Infections and infestations) | 0 | 1
Infection (Infections and infestations) | 1 | 0
Localised infection (Infections and infestations) | 0 | 2
Lower respiratory tract infection (Infections and infestations) | 0 | 4
Lung abscess (Infections and infestations) | 0 | 1
Lung infection (Infections and infestations) | 7 | 13
Neutropenic sepsis (Infections and infestations) | 1 | 1
Osteomyelitis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 20 | 44
Pneumonia bacterial (Infections and infestations) | 1 | 6
Respiratory tract infection (Infections and infestations) | 4 | 6
Sepsis (Infections and infestations) | 9 | 15
Septic encephalopathy (Infections and infestations) | 0 | 1
Septic shock (Infections and infestations) | 1 | 3
Staphylococcal infection (Infections and infestations) | 1 | 0
Superinfection viral (Infections and infestations) | 1 | 0
Tracheitis (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 2 | 1
Urinary tract infection (Infections and infestations) | 4 | 6
Urinary tract infection bacterial (Infections and infestations) | 2 | 1
Fall (Injury, poisoning and procedural complications) | 2 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 1 | 1
Fracture (Injury, poisoning and procedural complications) | 0 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 1 | 0
Injury (Injury, poisoning and procedural complications) | 1 | 1
Laceration (Injury, poisoning and procedural complications) | 1 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 1
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1
Nerve root injury lumbar (Injury, poisoning and procedural complications) | 0 | 1
Poisoning (Injury, poisoning and procedural complications) | 2 | 0
Procedural pneumothorax (Injury, poisoning and procedural complications) | 0 | 1
Radiation dysphagia (Injury, poisoning and procedural complications) | 1 | 0
Radiation pneumonitis (Injury, poisoning and procedural complications) | 0 | 2
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 0
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 1
Blood albumin abnormal (Investigations) | 0 | 1
Blood bilirubin increased (Investigations) | 0 | 1
Blood lactate dehydrogenase increased (Investigations) | 0 | 1
Blood pressure increased (Investigations) | 0 | 1
Eastern Cooperative Oncology Group performance status worsened (Investigations) | 0 | 1
Ejection fraction decreased (Investigations) | 0 | 1
Haemoglobin abnormal (Investigations) | 0 | 1
Haemoglobin decreased (Investigations) | 1 | 2
Liver function test abnormal (Investigations) | 0 | 2
Neutrophil count decreased (Investigations) | 0 | 1
Oxygen saturation decreased (Investigations) | 0 | 1
Platelet count decreased (Investigations) | 6 | 6
Salmonella test positive (Investigations) | 0 | 1
Transaminases increased (Investigations) | 0 | 1
White blood cell count decreased (Investigations) | 1 | 2
White blood cell count increased (Investigations) | 0 | 1
Acidosis (Metabolism and nutrition disorders) | 1 | 0
Cachexia (Metabolism and nutrition disorders) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 7
Dehydration (Metabolism and nutrition disorders) | 5 | 6
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 | 0
Electrolyte imbalance (Metabolism and nutrition disorders) | 2 | 2
Failure to thrive (Metabolism and nutrition disorders) | 1 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 4 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 1 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 5
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 2
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 3 | 2
Hypophagia (Metabolism and nutrition disorders) | 0 | 1
Hypoproteinaemia (Metabolism and nutrition disorders) | 1 | 1
Hypovolaemia (Metabolism and nutrition disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 3
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 | 2
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 | 1
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Lung adenocarcinoma stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Metastases to adrenals (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 3
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cerebellar infarction (Nervous system disorders) | 1 | 0
Cerebral haemorrhage (Nervous system disorders) | 0 | 1
Cerebral infarction (Nervous system disorders) | 0 | 4
Cerebral ischaemia (Nervous system disorders) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 1 | 4
Cognitive disorder (Nervous system disorders) | 0 | 1
Coma (Nervous system disorders) | 1 | 0
Dementia (Nervous system disorders) | 1 | 0
Depressed level of consciousness (Nervous system disorders) | 0 | 1
Diabetic neuropathy (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0
Encephalopathy (Nervous system disorders) | 2 | 1
Epilepsy (Nervous system disorders) | 2 | 1
Facial nerve disorder (Nervous system disorders) | 0 | 1
Haemorrhage intracranial (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 1 | 2
Hemiparesis (Nervous system disorders) | 0 | 1
Hemiplegia (Nervous system disorders) | 0 | 2
Hydrocephalus (Nervous system disorders) | 1 | 1
Hypoaesthesia (Nervous system disorders) | 0 | 1
Ischaemic stroke (Nervous system disorders) | 0 | 1
Lethargy (Nervous system disorders) | 0 | 2
Loss of consciousness (Nervous system disorders) | 0 | 1
Paraesthesia (Nervous system disorders) | 0 | 1
Paraplegia (Nervous system disorders) | 1 | 1
Partial seizures (Nervous system disorders) | 0 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 0
Presyncope (Nervous system disorders) | 1 | 0
Seizure (Nervous system disorders) | 2 | 4
Somnolence (Nervous system disorders) | 1 | 0
Stroke in evolution (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 1 | 1
Thrombotic cerebral infarction (Nervous system disorders) | 1 | 1
Thrombotic stroke (Nervous system disorders) | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 4
Unresponsive to stimuli (Nervous system disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 1 | 0
Completed suicide (Psychiatric disorders) | 1 | 0
Confusional state (Psychiatric disorders) | 0 | 1
Delirium (Psychiatric disorders) | 0 | 1
Depression (Psychiatric disorders) | 1 | 0
Disorientation (Psychiatric disorders) | 0 | 2
Mental status changes (Psychiatric disorders) | 1 | 1
Psychotic disorder (Psychiatric disorders) | 0 | 2
Acute kidney injury (Renal and urinary disorders) | 4 | 12
Azotaemia (Renal and urinary disorders) | 1 | 0
Chronic kidney disease (Renal and urinary disorders) | 0 | 1
Haematuria (Renal and urinary disorders) | 0 | 2
Obstructive uropathy (Renal and urinary disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 2 | 5
Urinary retention (Renal and urinary disorders) | 0 | 2
Vesical fistula (Renal and urinary disorders) | 0 | 1
Pelvic pain (Reproductive system and breast disorders) | 0 | 1
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 9
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Bronchial haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 4
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 26 | 31
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Emphysema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 3 | 14
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Oesophagobronchial fistula (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Painful respiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 12 | 6
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 4
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Pulmonary artery thrombosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 6 | 20
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 2 | 5
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory acidosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory depression (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 13 | 24
Peau d'orange (Skin and subcutaneous tissue disorders) | 0 | 1
Lymphadenectomy (Surgical and medical procedures) | 0 | 1
Thyroidectomy (Surgical and medical procedures) | 0 | 1
Accelerated hypertension (Vascular disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 3 | 11
Extremity necrosis (Vascular disorders) | 0 | 1
Hypertension (Vascular disorders) | 0 | 3
Hypotension (Vascular disorders) | 6 | 3
Hypovolaemic shock (Vascular disorders) | 1 | 1
Peripheral artery stenosis (Vascular disorders) | 0 | 1
Peripheral artery thrombosis (Vascular disorders) | 1 | 1
Peripheral embolism (Vascular disorders) | 1 | 0
Peripheral ischaemia (Vascular disorders) | 0 | 2
Superior vena cava occlusion (Vascular disorders) | 1 | 0
Superior vena cava syndrome (Vascular disorders) | 0 | 1
Thrombosis (Vascular disorders) | 0 | 1
Varicose ulceration (Vascular disorders) | 0 | 1
Vascular occlusion (Vascular disorders) | 0 | 1
Venous thrombosis limb (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=833) | Darbepoetin Alfa (N=1685)
Agranulocytosis (Blood and lymphatic system disorders) | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 244 | 451
Anaemia megaloblastic (Blood and lymphatic system disorders) | 0 | 1
Autoimmune haemolytic anaemia (Blood and lymphatic system disorders) | 0 | 1
Bandaemia (Blood and lymphatic system disorders) | 0 | 1
Bicytopenia (Blood and lymphatic system disorders) | 0 | 1
Bone marrow failure (Blood and lymphatic system disorders) | 16 | 39
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 | 0
Erythropenia (Blood and lymphatic system disorders) | 2 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 4
Granulocytopenia (Blood and lymphatic system disorders) | 3 | 11
Haematotoxicity (Blood and lymphatic system disorders) | 0 | 1
Haemolytic anaemia (Blood and lymphatic system disorders) | 1 | 0
Hypercoagulation (Blood and lymphatic system disorders) | 0 | 1
Increased tendency to bruise (Blood and lymphatic system disorders) | 0 | 1
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 4
Leukocytosis (Blood and lymphatic system disorders) | 5 | 11
Leukopenia (Blood and lymphatic system disorders) | 40 | 101
Lymph node pain (Blood and lymphatic system disorders) | 0 | 1
Lymphadenitis (Blood and lymphatic system disorders) | 0 | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 2
Lymphopenia (Blood and lymphatic system disorders) | 1 | 1
Neutropenia (Blood and lymphatic system disorders) | 79 | 202
Neutrophilia (Blood and lymphatic system disorders) | 1 | 1
Pancytopenia (Blood and lymphatic system disorders) | 2 | 4
Platelet disorder (Blood and lymphatic system disorders) | 2 | 4
Platelet production decreased (Blood and lymphatic system disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 66 | 156
Thrombocytopenia neonatal (Blood and lymphatic system disorders) | 0 | 1
Thrombocytosis (Blood and lymphatic system disorders) | 1 | 7
Acute coronary syndrome (Cardiac disorders) | 1 | 1
Angina pectoris (Cardiac disorders) | 1 | 3
Angina unstable (Cardiac disorders) | 1 | 0
Arrhythmia (Cardiac disorders) | 2 | 2
Arrhythmia supraventricular (Cardiac disorders) | 0 | 1
Arteriosclerosis coronary artery (Cardiac disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 2 | 2
Atrial tachycardia (Cardiac disorders) | 0 | 3
Cardiac discomfort (Cardiac disorders) | 0 | 1
Cardiac disorder (Cardiac disorders) | 0 | 1
Cardiac failure (Cardiac disorders) | 2 | 1
Cardiac failure congestive (Cardiac disorders) | 0 | 1
Cardiomyopathy (Cardiac disorders) | 0 | 1
Congestive cardiomyopathy (Cardiac disorders) | 0 | 1
Cyanosis (Cardiac disorders) | 0 | 2
Metabolic cardiomyopathy (Cardiac disorders) | 0 | 2
Myocardial infarction (Cardiac disorders) | 0 | 1
Myocardial ischaemia (Cardiac disorders) | 1 | 1
Palpitations (Cardiac disorders) | 2 | 4
Pericardial effusion (Cardiac disorders) | 1 | 0
Pericarditis (Cardiac disorders) | 0 | 1
Sinus arrhythmia (Cardiac disorders) | 1 | 0
Sinus tachycardia (Cardiac disorders) | 1 | 5
Supraventricular extrasystoles (Cardiac disorders) | 2 | 3
Supraventricular tachycardia (Cardiac disorders) | 1 | 0
Tachycardia (Cardiac disorders) | 7 | 10
Aplasia (Congenital, familial and genetic disorders) | 1 | 0
Deafness (Ear and labyrinth disorders) | 1 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 1
Hypoacusis (Ear and labyrinth disorders) | 0 | 4
Otorrhoea (Ear and labyrinth disorders) | 1 | 0
Tinnitus (Ear and labyrinth disorders) | 4 | 3
Vertigo (Ear and labyrinth disorders) | 4 | 5
Goitre (Endocrine disorders) | 1 | 0
Hypercalcaemia of malignancy (Endocrine disorders) | 0 | 1
Hyperthyroidism (Endocrine disorders) | 1 | 1
Thyroid dysfunction in pregnancy (Endocrine disorders) | 0 | 1
Asthenopia (Eye disorders) | 1 | 0
Blindness (Eye disorders) | 0 | 1
Blindness unilateral (Eye disorders) | 0 | 1
Cataract (Eye disorders) | 1 | 1
Conjunctival haemorrhage (Eye disorders) | 1 | 1
Conjunctival pallor (Eye disorders) | 0 | 1
Diplopia (Eye disorders) | 1 | 1
Dry eye (Eye disorders) | 1 | 3
Eye disorder (Eye disorders) | 2 | 0
Eye irritation (Eye disorders) | 0 | 2
Eye pain (Eye disorders) | 0 | 3
Eyelid margin crusting (Eye disorders) | 1 | 0
Eyelid oedema (Eye disorders) | 0 | 3
Glaucoma (Eye disorders) | 0 | 1
Keratitis (Eye disorders) | 0 | 1
Lacrimation increased (Eye disorders) | 5 | 7
Ocular hyperaemia (Eye disorders) | 0 | 1
Photophobia (Eye disorders) | 0 | 2
Pupils unequal (Eye disorders) | 1 | 0
Ulcerative keratitis (Eye disorders) | 1 | 0
Vision blurred (Eye disorders) | 3 | 3
Visual impairment (Eye disorders) | 0 | 1
Abdominal discomfort (Gastrointestinal disorders) | 3 | 6
Abdominal distension (Gastrointestinal disorders) | 8 | 9
Abdominal pain (Gastrointestinal disorders) | 18 | 50
Abdominal pain lower (Gastrointestinal disorders) | 2 | 5
Abdominal pain upper (Gastrointestinal disorders) | 15 | 17
Abdominal tenderness (Gastrointestinal disorders) | 2 | 0
Acute abdomen (Gastrointestinal disorders) | 1 | 0
Anal inflammation (Gastrointestinal disorders) | 1 | 0
Ascites (Gastrointestinal disorders) | 2 | 2
Chronic gastritis (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 56 | 106
Dental caries (Gastrointestinal disorders) | 0 | 2
Diarrhoea (Gastrointestinal disorders) | 46 | 106
Diverticulum intestinal (Gastrointestinal disorders) | 0 | 1
Dry mouth (Gastrointestinal disorders) | 1 | 1
Duodenitis (Gastrointestinal disorders) | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 5 | 12
Dysphagia (Gastrointestinal disorders) | 5 | 16
Enteritis (Gastrointestinal disorders) | 1 | 0
Epigastric discomfort (Gastrointestinal disorders) | 0 | 2
Faeces hard (Gastrointestinal disorders) | 0 | 1
Flatulence (Gastrointestinal disorders) | 1 | 3
Gastric polyps (Gastrointestinal disorders) | 0 | 1
Gastric ulcer (Gastrointestinal disorders) | 1 | 2
Gastritis (Gastrointestinal disorders) | 5 | 11
Gastrointestinal disorder (Gastrointestinal disorders) | 2 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 | 6
Gingival swelling (Gastrointestinal disorders) | 0 | 3
Glossitis (Gastrointestinal disorders) | 1 | 0
Glossodynia (Gastrointestinal disorders) | 1 | 0
Haematemesis (Gastrointestinal disorders) | 0 | 1
Haematochezia (Gastrointestinal disorders) | 2 | 2
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 2 | 1
Haemorrhoids (Gastrointestinal disorders) | 3 | 1
Hyperchlorhydria (Gastrointestinal disorders) | 0 | 3
Ileus (Gastrointestinal disorders) | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 1
Intestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Irritable bowel syndrome (Gastrointestinal disorders) | 0 | 1
Lip dry (Gastrointestinal disorders) | 0 | 1
Lip swelling (Gastrointestinal disorders) | 0 | 1
Melaena (Gastrointestinal disorders) | 1 | 0
Mouth ulceration (Gastrointestinal disorders) | 3 | 7
Nausea (Gastrointestinal disorders) | 101 | 187
Odynophagia (Gastrointestinal disorders) | 1 | 5
Oesophageal stenosis (Gastrointestinal disorders) | 1 | 0
Oesophagitis (Gastrointestinal disorders) | 2 | 2
Oral disorder (Gastrointestinal disorders) | 0 | 1
Oral pain (Gastrointestinal disorders) | 0 | 2
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 2
Rectal ulcer (Gastrointestinal disorders) | 0 | 1
Regurgitation (Gastrointestinal disorders) | 0 | 1
Retching (Gastrointestinal disorders) | 1 | 2
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Stomatitis (Gastrointestinal disorders) | 6 | 20
Tooth loss (Gastrointestinal disorders) | 0 | 1
Toothache (Gastrointestinal disorders) | 0 | 3
Vomiting (Gastrointestinal disorders) | 57 | 118
Adverse drug reaction (General disorders) | 0 | 3
Asthenia (General disorders) | 92 | 158
Axillary pain (General disorders) | 0 | 2
Catheter site haemorrhage (General disorders) | 1 | 0
Catheter site pain (General disorders) | 1 | 3
Chest discomfort (General disorders) | 2 | 5
Chest pain (General disorders) | 30 | 52
Chills (General disorders) | 5 | 9
Complication associated with device (General disorders) | 1 | 1
Extravasation (General disorders) | 0 | 1
Face oedema (General disorders) | 2 | 5
Facial pain (General disorders) | 1 | 1
Fatigue (General disorders) | 69 | 117
Feeling abnormal (General disorders) | 0 | 1
Feeling cold (General disorders) | 0 | 1
Gait disturbance (General disorders) | 1 | 4
General physical health deterioration (General disorders) | 0 | 2
Generalised oedema (General disorders) | 0 | 2
Gravitational oedema (General disorders) | 0 | 1
Hyperthermia (General disorders) | 1 | 2
Implant site pain (General disorders) | 0 | 1
Inflammation (General disorders) | 1 | 3
Influenza like illness (General disorders) | 2 | 3
Infusion site extravasation (General disorders) | 0 | 1
Injection site haematoma (General disorders) | 0 | 1
Injection site phlebitis (General disorders) | 0 | 1
Injection site reaction (General disorders) | 0 | 1
Local swelling (General disorders) | 0 | 3
Localised oedema (General disorders) | 1 | 2
Malaise (General disorders) | 6 | 14
Mass (General disorders) | 0 | 1
Mucosal inflammation (General disorders) | 8 | 7
Mucous membrane disorder (General disorders) | 0 | 1
Non-cardiac chest pain (General disorders) | 7 | 23
Oedema (General disorders) | 7 | 10
Oedema peripheral (General disorders) | 30 | 50
Pain (General disorders) | 18 | 41
Performance status decreased (General disorders) | 1 | 1
Peripheral swelling (General disorders) | 5 | 5
Pyrexia (General disorders) | 57 | 110
Temperature intolerance (General disorders) | 0 | 3
Vessel puncture site pain (General disorders) | 1 | 0
Vessel puncture site swelling (General disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 1
Chronic hepatic failure (Hepatobiliary disorders) | 0 | 3
Drug-induced liver injury (Hepatobiliary disorders) | 0 | 1
Gallbladder polyp (Hepatobiliary disorders) | 1 | 0
Hepatic cyst (Hepatobiliary disorders) | 0 | 2
Hepatic failure (Hepatobiliary disorders) | 0 | 1
Hepatic function abnormal (Hepatobiliary disorders) | 4 | 9
Hepatic lesion (Hepatobiliary disorders) | 1 | 0
Hepatic pain (Hepatobiliary disorders) | 1 | 1
Hepatic steatosis (Hepatobiliary disorders) | 1 | 1
Hepatotoxicity (Hepatobiliary disorders) | 0 | 2
Hyperbilirubinaemia (Hepatobiliary disorders) | 2 | 2
Hyperplastic cholecystopathy (Hepatobiliary disorders) | 0 | 1
Liver disorder (Hepatobiliary disorders) | 0 | 1
Liver injury (Hepatobiliary disorders) | 3 | 4
Ocular icterus (Hepatobiliary disorders) | 0 | 1
Anaphylactic reaction (Immune system disorders) | 0 | 1
Contrast media allergy (Immune system disorders) | 0 | 1
Drug hypersensitivity (Immune system disorders) | 5 | 2
Hypersensitivity (Immune system disorders) | 1 | 8
Immune system disorder (Immune system disorders) | 1 | 0
Immunodeficiency (Immune system disorders) | 0 | 1
Iodine allergy (Immune system disorders) | 0 | 1
Seasonal allergy (Immune system disorders) | 1 | 3
Abdominal wall infection (Infections and infestations) | 0 | 1
Alveolar osteitis (Infections and infestations) | 0 | 1
Amoebiasis (Infections and infestations) | 1 | 0
Anorectal cellulitis (Infections and infestations) | 1 | 0
Bacterial infection (Infections and infestations) | 1 | 0
Balanoposthitis infective (Infections and infestations) | 1 | 0
Bronchiolitis (Infections and infestations) | 0 | 1
Bronchitis (Infections and infestations) | 7 | 18
Bronchitis bacterial (Infections and infestations) | 1 | 0
Candida infection (Infections and infestations) | 1 | 2
Catheter site cellulitis (Infections and infestations) | 1 | 2
Cellulitis (Infections and infestations) | 2 | 5
Chikungunya virus infection (Infections and infestations) | 1 | 0
Clostridium difficile colitis (Infections and infestations) | 1 | 0
Conjunctivitis (Infections and infestations) | 3 | 4
Cystitis (Infections and infestations) | 1 | 2
Device related infection (Infections and infestations) | 0 | 4
Erysipelas (Infections and infestations) | 0 | 2
Eye infection (Infections and infestations) | 0 | 1
Febrile infection (Infections and infestations) | 1 | 1
Folliculitis (Infections and infestations) | 1 | 0
Fungal infection (Infections and infestations) | 2 | 2
Fungal skin infection (Infections and infestations) | 0 | 1
Furuncle (Infections and infestations) | 1 | 2
Gastroenteritis (Infections and infestations) | 1 | 3
Gastroenteritis viral (Infections and infestations) | 0 | 1
Gastrointestinal infection (Infections and infestations) | 0 | 1
Hepatitis B (Infections and infestations) | 2 | 2
Herpes dermatitis (Infections and infestations) | 0 | 1
Herpes simplex (Infections and infestations) | 0 | 1
Herpes virus infection (Infections and infestations) | 0 | 1
Herpes zoster (Infections and infestations) | 3 | 7
Infected bite (Infections and infestations) | 0 | 1
Infection (Infections and infestations) | 3 | 4
Influenza (Infections and infestations) | 5 | 8
Kidney infection (Infections and infestations) | 1 | 0
Localised infection (Infections and infestations) | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 1 | 6
Lung infection (Infections and infestations) | 6 | 12
Mastoiditis (Infections and infestations) | 0 | 2
Meningoencephalitis bacterial (Infections and infestations) | 0 | 1
Mucosal infection (Infections and infestations) | 0 | 1
Nasopharyngitis (Infections and infestations) | 1 | 1
Oesophageal candidiasis (Infections and infestations) | 0 | 1
Onychomycosis (Infections and infestations) | 0 | 1
Oral candidiasis (Infections and infestations) | 2 | 7
Oral fungal infection (Infections and infestations) | 1 | 1
Oral herpes (Infections and infestations) | 1 | 3
Oral infection (Infections and infestations) | 0 | 1
Orchitis (Infections and infestations) | 1 | 0
Oropharyngeal candidiasis (Infections and infestations) | 0 | 2
Paronychia (Infections and infestations) | 0 | 2
Penile infection (Infections and infestations) | 1 | 0
Pharyngitis (Infections and infestations) | 3 | 3
Pneumonia (Infections and infestations) | 13 | 26
Pneumonia bacterial (Infections and infestations) | 1 | 1
Post procedural infection (Infections and infestations) | 1 | 0
Rash pustular (Infections and infestations) | 0 | 1
Respiratory tract infection (Infections and infestations) | 3 | 9
Respiratory tract infection viral (Infections and infestations) | 5 | 5
Rhinitis (Infections and infestations) | 2 | 3
Sepsis (Infections and infestations) | 0 | 2
Sinusitis (Infections and infestations) | 1 | 4
Skin infection (Infections and infestations) | 1 | 0
Sputum purulent (Infections and infestations) | 1 | 0
Staphylococcal infection (Infections and infestations) | 0 | 1
Strongyloidiasis (Infections and infestations) | 0 | 1
Tinea cruris (Infections and infestations) | 0 | 1
Tonsillitis (Infections and infestations) | 0 | 1
Tooth infection (Infections and infestations) | 0 | 2
Tracheitis (Infections and infestations) | 0 | 1
Tracheobronchitis (Infections and infestations) | 3 | 2
Upper respiratory tract infection (Infections and infestations) | 14 | 33
Urinary tract infection (Infections and infestations) | 14 | 27
Urinary tract infection fungal (Infections and infestations) | 0 | 1
Viral infection (Infections and infestations) | 2 | 1
Viral upper respiratory tract infection (Infections and infestations) | 6 | 8
Vulvovaginal mycotic infection (Infections and infestations) | 1 | 0
Wound infection (Infections and infestations) | 0 | 1
Airway complication of anaesthesia (Injury, poisoning and procedural complications) | 0 | 1
Animal scratch (Injury, poisoning and procedural complications) | 0 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 1
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 1
Chemical poisoning (Injury, poisoning and procedural complications) | 0 | 1
Clavicle fracture (Injury, poisoning and procedural complications) | 0 | 1
Concussion (Injury, poisoning and procedural complications) | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 5 | 6
Fall (Injury, poisoning and procedural complications) | 3 | 7
Fracture (Injury, poisoning and procedural complications) | 0 | 2
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 3
Laceration (Injury, poisoning and procedural complications) | 2 | 3
Limb injury (Injury, poisoning and procedural complications) | 0 | 1
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1
Overdose (Injury, poisoning and procedural complications) | 0 | 1
Poisoning (Injury, poisoning and procedural complications) | 4 | 4
Post procedural fistula (Injury, poisoning and procedural complications) | 0 | 1
Procedural pain (Injury, poisoning and procedural complications) | 0 | 1
Radiation oesophagitis (Injury, poisoning and procedural complications) | 0 | 2
Radiation pneumonitis (Injury, poisoning and procedural complications) | 1 | 0
Radiation skin injury (Injury, poisoning and procedural complications) | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 1 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 1 | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 1
Tooth fracture (Injury, poisoning and procedural complications) | 0 | 1
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 | 1
Upper limb fracture (Injury, poisoning and procedural complications) | 1 | 0
Wound (Injury, poisoning and procedural complications) | 0 | 1
Wound complication (Injury, poisoning and procedural complications) | 1 | 1
Alanine aminotransferase (Investigations) | 0 | 2
Alanine aminotransferase decreased (Investigations) | 0 | 2
Alanine aminotransferase increased (Investigations) | 26 | 43
Albumin CSF decreased (Investigations) | 0 | 1
Alpha hydroxybutyrate dehydrogenase increased (Investigations) | 0 | 1
Antineutrophil cytoplasmic antibody decreased (Investigations) | 0 | 1
Aspartate aminotransferase decreased (Investigations) | 0 | 1
Aspartate aminotransferase increased (Investigations) | 21 | 38
Aspiration pleural cavity (Investigations) | 0 | 1
Biopsy pleura (Investigations) | 1 | 0
Blood albumin decreased (Investigations) | 5 | 7
Blood alkaline phosphatase increased (Investigations) | 7 | 20
Blood bicarbonate decreased (Investigations) | 1 | 1
Blood bicarbonate increased (Investigations) | 1 | 0
Blood bilirubin increased (Investigations) | 0 | 2
Blood bilirubin unconjugated increased (Investigations) | 0 | 1
Blood calcitonin increased (Investigations) | 1 | 1
Blood calcium decreased (Investigations) | 1 | 1
Blood chloride decreased (Investigations) | 1 | 2
Blood chloride increased (Investigations) | 0 | 1
Blood cholesterol increased (Investigations) | 0 | 2
Blood creatine (Investigations) | 0 | 1
Blood creatine abnormal (Investigations) | 1 | 2
Blood creatine increased (Investigations) | 0 | 6
Blood creatine phosphokinase MB increased (Investigations) | 0 | 1
Blood creatinine (Investigations) | 0 | 1
Blood creatinine increased (Investigations) | 16 | 27
Blood glucose increased (Investigations) | 5 | 6
Blood iron abnormal (Investigations) | 0 | 1
Blood iron decreased (Investigations) | 0 | 3
Blood lactate dehydrogenase increased (Investigations) | 8 | 13
Blood potassium decreased (Investigations) | 2 | 6
Blood pressure increased (Investigations) | 2 | 2
Blood pressure systolic increased (Investigations) | 1 | 0
Blood testosterone decreased (Investigations) | 0 | 1
Blood thyroid stimulating hormone decreased (Investigations) | 1 | 0
Blood triglycerides increased (Investigations) | 1 | 0
Blood urea decreased (Investigations) | 1 | 1
Blood urea increased (Investigations) | 6 | 10
Blood uric acid increased (Investigations) | 2 | 4
Body temperature increased (Investigations) | 3 | 1
Brain natriuretic peptide increased (Investigations) | 0 | 1
Breath sounds abnormal (Investigations) | 2 | 1
C-reactive protein increased (Investigations) | 0 | 2
Creatinine renal clearance decreased (Investigations) | 2 | 3
Creatinine renal clearance increased (Investigations) | 0 | 1
Eastern Cooperative Oncology Group performance status worsened (Investigations) | 1 | 4
Electrocardiogram QT prolonged (Investigations) | 0 | 2
Fibrin D dimer increased (Investigations) | 0 | 2
Fibrin degradation products increased (Investigations) | 0 | 1
Gamma-glutamyltransferase (Investigations) | 0 | 1
Gamma-glutamyltransferase decreased (Investigations) | 0 | 1
Gamma-glutamyltransferase increased (Investigations) | 10 | 22
Gastric pH decreased (Investigations) | 1 | 0
General physical condition abnormal (Investigations) | 0 | 1
Globulins decreased (Investigations) | 0 | 1
Glomerular filtration rate decreased (Investigations) | 0 | 1
Glucose tolerance decreased (Investigations) | 1 | 0
Glucose urine present (Investigations) | 0 | 1
Glycosylated haemoglobin increased (Investigations) | 1 | 0
Granulocyte count decreased (Investigations) | 2 | 9
Haematocrit decreased (Investigations) | 1 | 0
Haemoglobin decreased (Investigations) | 10 | 8
Heart rate increased (Investigations) | 2 | 1
Hepatic enzyme increased (Investigations) | 1 | 2
Human epidermal growth factor receptor decreased (Investigations) | 1 | 0
International normalised ratio increased (Investigations) | 1 | 1
Iron binding capacity total decreased (Investigations) | 0 | 1
Iron binding capacity unsaturated decreased (Investigations) | 0 | 1
Laboratory test abnormal (Investigations) | 1 | 0
Liver function test abnormal (Investigations) | 1 | 10
Liver function test increased (Investigations) | 0 | 1
Lymphocyte count abnormal (Investigations) | 0 | 1
Lymphocyte count decreased (Investigations) | 5 | 15
Lymphocyte count increased (Investigations) | 0 | 1
Mean cell volume increased (Investigations) | 1 | 0
Monocyte percentage increased (Investigations) | 0 | 1
Myoglobin blood increased (Investigations) | 0 | 1
Neutrophil count (Investigations) | 1 | 1
Neutrophil count abnormal (Investigations) | 1 | 1
Neutrophil count decreased (Investigations) | 47 | 95
Neutrophil count increased (Investigations) | 0 | 5
Neutrophil percentage increased (Investigations) | 0 | 2
PCO2 decreased (Investigations) | 0 | 1
Platelet adhesiveness decreased (Investigations) | 1 | 0
Platelet adhesiveness increased (Investigations) | 0 | 1
Platelet count abnormal (Investigations) | 0 | 1
Platelet count decreased (Investigations) | 66 | 130
Platelet count increased (Investigations) | 2 | 3
Protein total decreased (Investigations) | 1 | 2
Protein total increased (Investigations) | 1 | 0
Protein urine present (Investigations) | 1 | 0
Respiratory rate decreased (Investigations) | 0 | 1
Serum ferritin decreased (Investigations) | 0 | 1
Serum ferritin increased (Investigations) | 1 | 1
Transaminases increased (Investigations) | 1 | 0
Troponin I increased (Investigations) | 0 | 1
Troponin increased (Investigations) | 0 | 1
Urine output decreased (Investigations) | 1 | 1
Vitamin D decreased (Investigations) | 0 | 1
Weight decreased (Investigations) | 24 | 53
Weight increased (Investigations) | 4 | 4
White blood cell count (Investigations) | 1 | 1
White blood cell count decreased (Investigations) | 64 | 138
White blood cell count increased (Investigations) | 3 | 7
White blood cells urine positive (Investigations) | 0 | 1
Acidosis (Metabolism and nutrition disorders) | 0 | 1
Cachexia (Metabolism and nutrition disorders) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 63 | 134
Dehydration (Metabolism and nutrition disorders) | 14 | 37
Diabetes mellitus (Metabolism and nutrition disorders) | 4 | 1
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 2 | 0
Dyslipidaemia (Metabolism and nutrition disorders) | 0 | 1
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 | 1
Fluid retention (Metabolism and nutrition disorders) | 1 | 0
Glucose tolerance impaired (Metabolism and nutrition disorders) | 1 | 0
Gout (Metabolism and nutrition disorders) | 2 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 5 | 4
Hyperchloraemia (Metabolism and nutrition disorders) | 0 | 1
Hypercholesterolaemia (Metabolism and nutrition disorders) | 3 | 1
Hypercreatininaemia (Metabolism and nutrition disorders) | 2 | 4
Hyperglycaemia (Metabolism and nutrition disorders) | 14 | 32
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 7
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 | 1
Hypernatraemia (Metabolism and nutrition disorders) | 1 | 2
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 | 1
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 | 3
Hyperuricaemia (Metabolism and nutrition disorders) | 2 | 8
Hypoalbuminaemia (Metabolism and nutrition disorders) | 16 | 47
Hypocalcaemia (Metabolism and nutrition disorders) | 11 | 25
Hypochloraemia (Metabolism and nutrition disorders) | 2 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 4 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 36 | 53
Hypomagnesaemia (Metabolism and nutrition disorders) | 10 | 9
Hyponatraemia (Metabolism and nutrition disorders) | 12 | 25
Hypophagia (Metabolism and nutrition disorders) | 1 | 2
Hypophosphataemia (Metabolism and nutrition disorders) | 3 | 0
Hypoproteinaemia (Metabolism and nutrition disorders) | 11 | 9
Hypovolaemia (Metabolism and nutrition disorders) | 0 | 1
Iron deficiency (Metabolism and nutrition disorders) | 0 | 2
Iron overload (Metabolism and nutrition disorders) | 0 | 1
Malnutrition (Metabolism and nutrition disorders) | 1 | 4
Marasmus (Metabolism and nutrition disorders) | 1 | 0
Metabolic disorder (Metabolism and nutrition disorders) | 1 | 0
Protein deficiency (Metabolism and nutrition disorders) | 0 | 2
Tetany (Metabolism and nutrition disorders) | 0 | 1
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 | 1
Vitamin D deficiency (Metabolism and nutrition disorders) | 1 | 1
Weight loss poor (Metabolism and nutrition disorders) | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 21 | 32
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 35 | 65
Bone formation increased (Musculoskeletal and connective tissue disorders) | 1 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 10 | 30
Bursitis (Musculoskeletal and connective tissue disorders) | 1 | 1
Coccydynia (Musculoskeletal and connective tissue disorders) | 0 | 1
Connective tissue disorder (Musculoskeletal and connective tissue disorders) | 0 | 1
Exostosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Fistula (Musculoskeletal and connective tissue disorders) | 0 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 5
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Hypercreatinaemia (Musculoskeletal and connective tissue disorders) | 1 | 3
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 1 | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 2 | 1
Limb discomfort (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle fatigue (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 5 | 6
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 9 | 12
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 8 | 17
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 12 | 25
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 12 | 26
Neck pain (Musculoskeletal and connective tissue disorders) | 4 | 7
Osteolysis (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 22 | 57
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 2
Patellofemoral pain syndrome (Musculoskeletal and connective tissue disorders) | 1 | 1
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 | 1
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 1
Spinal pain (Musculoskeletal and connective tissue disorders) | 1 | 5
Synovial cyst (Musculoskeletal and connective tissue disorders) | 1 | 1
Trismus (Musculoskeletal and connective tissue disorders) | 1 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 8
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Paraneoplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 6
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Amnesia (Nervous system disorders) | 0 | 2
Anaesthesia (Nervous system disorders) | 0 | 1
Aphasia (Nervous system disorders) | 0 | 1
Aphonia (Nervous system disorders) | 0 | 1
Ataxia (Nervous system disorders) | 2 | 5
Burning sensation (Nervous system disorders) | 1 | 2
Central nervous system lesion (Nervous system disorders) | 1 | 0
Central pain syndrome (Nervous system disorders) | 0 | 1
Cerebral atrophy (Nervous system disorders) | 0 | 2
Cerebral infarction (Nervous system disorders) | 0 | 1
Cerebral ischaemia (Nervous system disorders) | 1 | 0
Cerebrovascular disorder (Nervous system disorders) | 1 | 0
Cervical radiculopathy (Nervous system disorders) | 0 | 1
Cognitive disorder (Nervous system disorders) | 1 | 2
Diabetic neuropathy (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 24 | 58
Dizziness postural (Nervous system disorders) | 0 | 2
Dysarthria (Nervous system disorders) | 1 | 1
Dysgeusia (Nervous system disorders) | 2 | 7
Dyskinesia (Nervous system disorders) | 0 | 2
Encephalopathy (Nervous system disorders) | 1 | 0
Epilepsy (Nervous system disorders) | 1 | 0
Facial paralysis (Nervous system disorders) | 0 | 1
Head discomfort (Nervous system disorders) | 0 | 2
Headache (Nervous system disorders) | 18 | 55
Hemiparesis (Nervous system disorders) | 2 | 4
Hemiplegia (Nervous system disorders) | 0 | 2
Hypoaesthesia (Nervous system disorders) | 13 | 21
Hypogeusia (Nervous system disorders) | 2 | 2
Intellectual disability (Nervous system disorders) | 0 | 1
Intercostal neuralgia (Nervous system disorders) | 1 | 0
Lethargy (Nervous system disorders) | 0 | 3
Loss of consciousness (Nervous system disorders) | 0 | 3
Migraine (Nervous system disorders) | 1 | 1
Monoparesis (Nervous system disorders) | 0 | 1
Nervous system disorder (Nervous system disorders) | 0 | 1
Neuralgia (Nervous system disorders) | 1 | 3
Neuropathy peripheral (Nervous system disorders) | 40 | 57
Paraesthesia (Nervous system disorders) | 14 | 26
Peripheral motor neuropathy (Nervous system disorders) | 3 | 4
Peripheral sensory neuropathy (Nervous system disorders) | 21 | 39
Polyneuropathy (Nervous system disorders) | 5 | 6
Poor quality sleep (Nervous system disorders) | 1 | 2
Presyncope (Nervous system disorders) | 0 | 1
Psychomotor hyperactivity (Nervous system disorders) | 0 | 2
Sciatica (Nervous system disorders) | 1 | 0
Seizure (Nervous system disorders) | 3 | 4
Sensory disturbance (Nervous system disorders) | 0 | 1
Somnolence (Nervous system disorders) | 1 | 4
Syncope (Nervous system disorders) | 3 | 10
Tremor (Nervous system disorders) | 2 | 4
Device leakage (Product Issues) | 0 | 1
Agitation (Psychiatric disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 9 | 18
Anxiety disorder (Psychiatric disorders) | 1 | 0
Anxiety disorder due to a general medical condition (Psychiatric disorders) | 0 | 1
Confusional state (Psychiatric disorders) | 4 | 6
Delirium (Psychiatric disorders) | 0 | 1
Depressed mood (Psychiatric disorders) | 2 | 0
Depression (Psychiatric disorders) | 8 | 11
Dysphoria (Psychiatric disorders) | 0 | 1
Flight of ideas (Psychiatric disorders) | 0 | 1
Hallucination (Psychiatric disorders) | 0 | 1
Hyposomnia (Psychiatric disorders) | 1 | 2
Initial insomnia (Psychiatric disorders) | 0 | 1
Insomnia (Psychiatric disorders) | 22 | 41
Insomnia related to another mental condition (Psychiatric disorders) | 0 | 1
Mental disorder (Psychiatric disorders) | 0 | 1
Mental status changes (Psychiatric disorders) | 0 | 2
Mood swings (Psychiatric disorders) | 1 | 0
Organic brain syndrome (Psychiatric disorders) | 1 | 0
Restlessness (Psychiatric disorders) | 1 | 0
Sleep disorder (Psychiatric disorders) | 3 | 1
Tic (Psychiatric disorders) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 3 | 5
Anuria (Renal and urinary disorders) | 0 | 1
Bladder dilatation (Renal and urinary disorders) | 1 | 0
Calculus bladder (Renal and urinary disorders) | 0 | 1
Chronic kidney disease (Renal and urinary disorders) | 1 | 1
Dysuria (Renal and urinary disorders) | 1 | 11
Glycosuria (Renal and urinary disorders) | 1 | 0
Haematuria (Renal and urinary disorders) | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 1
Nephropathy (Renal and urinary disorders) | 0 | 2
Nocturia (Renal and urinary disorders) | 0 | 1
Oliguria (Renal and urinary disorders) | 0 | 4
Pollakiuria (Renal and urinary disorders) | 3 | 2
Proteinuria (Renal and urinary disorders) | 2 | 2
Renal failure (Renal and urinary disorders) | 5 | 5
Renal impairment (Renal and urinary disorders) | 1 | 4
Renal pain (Renal and urinary disorders) | 0 | 3
Urinary hesitation (Renal and urinary disorders) | 1 | 1
Urinary incontinence (Renal and urinary disorders) | 0 | 4
Urinary retention (Renal and urinary disorders) | 3 | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 | 2
Breast mass (Reproductive system and breast disorders) | 0 | 1
Breast pain (Reproductive system and breast disorders) | 1 | 0
Breast swelling (Reproductive system and breast disorders) | 1 | 0
Menorrhagia (Reproductive system and breast disorders) | 0 | 1
Pelvic pain (Reproductive system and breast disorders) | 3 | 0
Postmenopausal haemorrhage (Reproductive system and breast disorders) | 0 | 1
Prostatitis (Reproductive system and breast disorders) | 0 | 1
Scrotal oedema (Reproductive system and breast disorders) | 0 | 1
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 1
Vulvovaginal pruritus (Reproductive system and breast disorders) | 1 | 0
Allergic respiratory symptom (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Apnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Bronchial haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 2 | 5
Bronchostenosis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 9
Cough (Respiratory, thoracic and mediastinal disorders) | 52 | 147
Dry throat (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 4 | 12
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 60 | 111
Dyspnoea at rest (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 8 | 21
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 11 | 31
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 24 | 42
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 | 7
Hypopnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Laryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 | 5
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Nasal mucosal ulcer (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 7 | 15
Orthopnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Paranasal sinus hypersecretion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pharyngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 4 | 8
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 15 | 31
Pulmonary arterial hypertension (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 7
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory tract haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 3 | 6
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 6
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Sputum discoloured (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Sputum retention (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Wheezing (Respiratory, thoracic and mediastinal disorders) | 2 | 4
Acne (Skin and subcutaneous tissue disorders) | 1 | 2
Actinic keratosis (Skin and subcutaneous tissue disorders) | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 70 | 125
Cold sweat (Skin and subcutaneous tissue disorders) | 0 | 1
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 4 | 4
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 1
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 1
Dermatitis bullous (Skin and subcutaneous tissue disorders) | 0 | 1
Drug eruption (Skin and subcutaneous tissue disorders) | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 4
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 | 4
Eczema (Skin and subcutaneous tissue disorders) | 1 | 1
Erythema (Skin and subcutaneous tissue disorders) | 5 | 4
Haemorrhage subcutaneous (Skin and subcutaneous tissue disorders) | 1 | 0
Hand dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 4
Ingrowing nail (Skin and subcutaneous tissue disorders) | 0 | 1
Nail discolouration (Skin and subcutaneous tissue disorders) | 0 | 1
Nail disorder (Skin and subcutaneous tissue disorders) | 2 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 3 | 2
Pain of skin (Skin and subcutaneous tissue disorders) | 0 | 1
Palmar erythema (Skin and subcutaneous tissue disorders) | 0 | 1
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 1
Petechiae (Skin and subcutaneous tissue disorders) | 1 | 3
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 | 1
Pigmentation disorder (Skin and subcutaneous tissue disorders) | 1 | 1
Plantar erythema (Skin and subcutaneous tissue disorders) | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 22
Pruritus allergic (Skin and subcutaneous tissue disorders) | 0 | 1
Pruritus generalised (Skin and subcutaneous tissue disorders) | 3 | 1
Purpura (Skin and subcutaneous tissue disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 14 | 25
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 1
Rash generalised (Skin and subcutaneous tissue disorders) | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 2
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 2
Skin discolouration (Skin and subcutaneous tissue disorders) | 0 | 1
Skin disorder (Skin and subcutaneous tissue disorders) | 1 | 0
Skin erosion (Skin and subcutaneous tissue disorders) | 0 | 1
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 | 1
Skin fissures (Skin and subcutaneous tissue disorders) | 0 | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 1
Skin mass (Skin and subcutaneous tissue disorders) | 0 | 1
Skin odour abnormal (Skin and subcutaneous tissue disorders) | 0 | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 2
Subcutaneous emphysema (Skin and subcutaneous tissue disorders) | 0 | 1
Swelling face (Skin and subcutaneous tissue disorders) | 3 | 2
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 1
Xeroderma (Skin and subcutaneous tissue disorders) | 0 | 1
Cataract operation (Surgical and medical procedures) | 1 | 0
Constipation prophylaxis (Surgical and medical procedures) | 0 | 1
Joint arthroplasty (Surgical and medical procedures) | 0 | 1
Leg amputation (Surgical and medical procedures) | 0 | 1
Pneumonolysis (Surgical and medical procedures) | 1 | 0
Reduction of increased intracranial pressure (Surgical and medical procedures) | 1 | 0
Angiopathy (Vascular disorders) | 1 | 0
Arterial disorder (Vascular disorders) | 1 | 0
Arteriosclerosis (Vascular disorders) | 0 | 3
Deep vein thrombosis (Vascular disorders) | 7 | 8
Diastolic hypertension (Vascular disorders) | 2 | 0
Embolism (Vascular disorders) | 0 | 1
Extremity necrosis (Vascular disorders) | 0 | 1
Flushing (Vascular disorders) | 0 | 4
Haematoma (Vascular disorders) | 1 | 2
Haemorrhage (Vascular disorders) | 1 | 1
Hot flush (Vascular disorders) | 2 | 1
Hypertension (Vascular disorders) | 21 | 35
Hypotension (Vascular disorders) | 6 | 11
Intermittent claudication (Vascular disorders) | 0 | 1
Orthostatic hypotension (Vascular disorders) | 1 | 0
Pallor (Vascular disorders) | 2 | 3
Pelvic venous thrombosis (Vascular disorders) | 0 | 1
Peripheral artery occlusion (Vascular disorders) | 0 | 1
Peripheral artery thrombosis (Vascular disorders) | 1 | 0
Peripheral venous disease (Vascular disorders) | 0 | 1
Phlebitis (Vascular disorders) | 1 | 5
Phlebitis superficial (Vascular disorders) | 1 | 0
Superior vena cava syndrome (Vascular disorders) | 2 | 3
Thrombophlebitis (Vascular disorders) | 0 | 3
Thrombophlebitis superficial (Vascular disorders) | 1 | 0
Thrombosis (Vascular disorders) | 0 | 5
Varicose vein (Vascular disorders) | 1 | 0
Vascular insufficiency (Vascular disorders) | 0 | 1
Vena cava thrombosis (Vascular disorders) | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.

DOCUMENTS (2):
  • Study Protocol (2012-11-13): https://cdn.clinicaltrials.gov/large-docs/64/NCT00858364/Prot_001.pdf
  • Statistical Analysis Plan (2017-09-14): https://cdn.clinicaltrials.gov/large-docs/64/NCT00858364/SAP_000.pdf